CLINICAL TRIAL: NCT01493700
Title: Effect of Heated Humidifier on the Body Temperature During Shouler Arthroscopy
Brief Title: Changes of Body Temperature During Shoulder Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Youn Yi Jo, Asistant professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: GIRBA 2612
Record Dates: First submitted 2011-12-08; First posted 2011-12-16 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Hypothermia
Keywords: heated circuit; body temperature
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Experimental): use routine respiratory circuit during mechanical ventilation of anesthetic machine during shoulder arthroscopy
  Interventions: Procedure: heated circuit
- electrically heated circuit (Active Comparator): use routine respiratory circuit during mechanical ventilation of anesthetic machine during shoulder arthroscopy
  Interventions: Procedure: control

INTERVENTIONS:
Procedure: heated circuit — use electrically heated respiratory circuit (set at 37oC)during mechanical ventilation of anesthetic machine during shoulder arthroscopy
  Other Names: heat circuit
  Arms: control
Procedure: control — use routine respiratory circuit during mechanical ventilation of anesthetic machine during shoulder arthroscopy
  Arms: electrically heated circuit

SUMMARY:
The purpose of this study is to compare the effect of electrically heated humidifier on the body temperature during shoulder arthroscopy.

DETAILED DESCRIPTION:
On the control group, use only routine anesthetic respiratory circuit for mechanical ventilation On the comparative group, use electrically heated humidifier for mechanical ventilation And compared the changes of body temperature durgin shoulder artheroscopy.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologist physical status 1 or 2
* 20-60 years old

Exclusion Criteria:

* body mass index over 30 kg/m2
* peripheral vascular disease
* uncontrolled cardiovascular disease

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
changes of body temperature | every 15 minutes from base line
  record the changes of esophageal and peripheral body temperature every 15 minutes from base line during shouler arthroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Cheon Lee, MD.PhD, Study Director — Gachon University Gil Medical Center
Locations (1):
- Kyung Cheon Lee, Incheon, South Korea

REFERENCES:
- [Result] Lee HK, Jang YH, Choi KW, Lee JH. The effect of electrically heated humidifier on the body temperature and blood loss in spinal surgery under general anesthesia. Korean J Anesthesiol. 2011 Aug;61(2):112-6. doi: 10.4097/kjae.2011.61.2.112. Epub 2011 Aug 23. PMID 21927679